CLINICAL TRIAL: NCT05650320
Title: A Multicenter, Randomized, Double-Blind, Vehicle-Controlled, Parallel-Group Clinical Trial to Demonstrate the Superiority of 0.3% and 1% OPA-15406 Ointment Versus Vehicle in Pediatric Subjects with Atopic Dermatitis
Brief Title: To Demonstrate the Superiority of IMP (0.3% and 1% OPA-15406 Ointment) Versus the Vehicle in Pediatric Patients with AD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 271-403-00013
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic | interventions — difamilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 0.3% OPA-15406 Ointment (Experimental): The 0.3% formulation of OPA-15406 ointment will be administered twice-daily (approximately 12 hours apart between morning and night administration) for 4 weeks. The amount of IMP (g) per dose is 10 g/m2 BSA and calculated.
  Interventions: Drug: 0.3% OPA-15406 Ointment
- 1% OPA-15406 Ointment (Experimental): The 1% formulation of OPA-15406 ointment will be administered twice-daily (approximately 12 hours apart between morning and night administration) for 4 weeks. The amount of IMP (g) per dose is 10 g/m2 BSA and calculated.
  Interventions: Drug: 1% OPA-15406 Ointment
- 0% OPA-15406 Vehicle (Placebo Comparator): The 0% formulation of OPA-15406 venicle will be administered twice-daily (approximately 12 hours apart between morning and night administration) for 4 weeks. The amount of IMP (g) per dose is 10 g/m2 BSA and calculated.
  Interventions: Other: 0% OPA-15406 vehicle

INTERVENTIONS:
Drug: 0.3% OPA-15406 Ointment — Twice-daily administration for 4 weeks.
  Arms: 0.3% OPA-15406 Ointment
Drug: 1% OPA-15406 Ointment — Twice-daily administration for 4 weeks.
  Arms: 1% OPA-15406 Ointment
Other: 0% OPA-15406 vehicle — Twice-daily administration for 4 weeks.
  Arms: 0% OPA-15406 Vehicle

SUMMARY:
A multicenter, randomized, double-blind, vehicle-controlled, parallel group trial to demonstrate the superiority of 0.3% and 1% OPA-15406 ointment to vehicle in pediatric subjects with AD. This trial consists of the 0.3% OPA-15406 group, the 1% OPA-15406 group, and the vehicle group.

DETAILED DESCRIPTION:
1. Screening period is defined as the interval between the day of obtaining informed consent and the day of the baseline visit (0-30 days). The investigator performs a screening examination after obtaining informed consent from the subject's legal guardian (and, if possible, after obtaining consent from the subject).
2. Assessment period (4 weeks double blind treatment period) is defined as the period between the day of baseline visit and the end of Week 4 visit (or the end of withdrawal visit). Subjects who meet the inclusion criteria and do not meet the exclusion criteria at the baseline visit will be assigned to receive 0.3% or 1% OPA-15406 ointment or comparator (vehicle [Placebo]). The allocated IMP will be administered to the treatment area from the day of baseline visit twice-daily for 4 weeks. After the baseline visit, examinations will be performed at Weeks 1, 2, and 4. If a subject discontinues the IMP administration between the day of baseline visit and the day of the Week 4 visit, a withdrawal visit will be performed for that subject.
3. Trial period(4 weeks double blind Treatment) The trial period for an individual subject is the period from the day of obtaining the written informed consent from the subject's legal guardian to the day of the Week 4 visit or withdrawal visit. For subjects who miss the Week 4 visit or withdrawal visit, the termination date, will be the date, as determined by the investigator, when the subject is withdrawn from the trial. The trial period does not include a follow-up period for AE.
4. 24 weeks, Open label, long term treatment period To be eligible for long term treatment, subjects must complete the randomized, double-blind treatment. Subjects must be judged by their investigators to have the potential for clinical benefit by longer-term exposure to OPA-15406, they can continue to receive 0.3% or 1% OPA-15406 open treatment for up to 24 weeks based on the inform consent of the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: Either male or female. Age: 2 to 14 years, inclusive (at time of obtaining informed consent) (only for 4 weeks double blind treatment).
2. Diagnosis of AD based on the criteria of Hanifin and Rajka (see Appendix 1).
3. Atopic dermatitis affecting ≥5% to ≤40% of BSA (excluding scalp) at the screening and baseline visit(only for 4 weeks double blind treatment).

Exclusion Criteria:

1. Subjects who defined as AD or contact dermatitis rapid deterioration, within 28 days prior to the baseline visit.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2024-07-21 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Success rate in Investigator's Global Assessment at Week 4 | 4 weeks
  Investigator's Global Assessment measures the severity of atopic dermatitis (0 = Clear; 1 = Almost clear; 2 = Mild disease; 3 = Moderate disease; 4 = Severe disease/Very severe disease) of clinical characteristics (erythema, infiltration, papulation, oozing, and crusting). A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by percentage of subjects with Investigator's Global Assessment score of 0 or 1 with improvement by at least 2 grades from baseline. Subjects with missing Investigator's Global Assessmen data will be handled as non-responders.

SECONDARY OUTCOMES:
Change from baseline in Investigator's Global Assessment at Week 4 | 4 weeks
  Investigator's Global Assessment measures the severity of atopic dermatitis (0 = Clear; 1 = Almost clear; 2 = Mild disease; 3 = Moderate disease; 4 = Severe disease/Very severe disease) of clinical characteristics (erythema, infiltration, papulation, oozing, and crusting). A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by the change from baseline in Investigator's Global Assessment at Week 4.
Success rate in Eczema Area and Severity Index 50 (improvement of ≥50% in Eczema Area and Severity Index) and at Week 4. | 4 weeks
  Eczema Area and Severity Index measures the severity of skin symptoms. The maximum Eczema Area and Severity Index score is 72 points. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by success rate in Eczema Area and Severity Index 50 (improvement of ≥50% in Eczema Area and Severity Index) and at Week 4.
Success rate in Eczema Area and Severity Index 75 (improvement of ≥75% in Eczema Area and Severity Index) and at Week 4. | 4 weeks
  Eczema Area and Severity Index measures the severity of skin symptoms. The maximum Eczema Area and Severity Index score is 72 points. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by the success rate in Eczema Area and Severity Index 75 (improvement of ≥75% in Eczema Area and Severity Index) at Week 4.
Eczema Area and Severity Index 90 (improvement of ≥90% in Eczema Area and Severity Index) at week 4 | 4 weeks
  Eczema Area and Severity Index measures the severity of skin symptoms. The maximum Eczema Area and Severity Index score is 72 points. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by success rate in Eczema Area and Severity Index 90 (improvement of ≥90% in Eczema Area and Severity Index) and at Week 4.
Change from baseline in the total score of Eczema Area and Severity Index and each clinical sign score at Week 4 | 4 weeks
  Eczema Area and Severity Index measures the severity of skin symptoms. The maximum Eczema Area and Severity Index score is 72 points. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by change from baseline in the total score of Eczema Area and Severity Index and each clinical sign score at Week 4.
Change from baseline in Verbal Rating Scale for Pruritus at Week 4 | 4 weeks
  The Verbal Rating Scale measures the intense pruritus in the past 24 hours following Verbal Rating Scale criteria( 0: None,1: Mild, 2: Moderate, 3: Severe). A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by Change from baseline in Verbal Rating Scale for Pruritus at Week 4
Change from baseline in Verbal Rating Scale for pruritus up to Day 7 | 7 Days
  The Verbal Rating Scale measures the intense pruritus in the past 24 hours following Verbal Rating Scale criteria( 0: None,1: Mild, 2: Moderate, 3: Severe). A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's/subjects' judgment.
  The efficacy is assessed by Change from baseline in Verbal Rating Scale for Pruritus up to day 7.
Change from baseline in the total score of Patient-Oriented Eczema Measure at Week 4 | 4 Weeks
  Eczema will be evaluated according to Patient-Oriented Eczema Measure .The subjects will answer 7 questions and describe their eczema. The investigator will confirm their responses and record the results in the source document and CRF. The total score of POEM is 28 points at the most. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by Change from baseline in the total score of Patient-Oriented Eczema Measure at Week 4
Change from baseline in the total affected Body Surface Area (percent) at Week 4 | 4 weeks
  The efficacy is assessed by change from baseline in the total affected Body Surface Area (percent) at Week 4.
Success rate in Investigator's Global Assessment | 24 Weeks
  Investigator's Global Assessment measures the severity of atopic dermatitis (0 = Clear; 1 = Almost clear; 2 = Mild disease; 3 = Moderate disease; 4 = Severe disease/Very severe disease) of clinical characteristics (erythema, infiltration, papulation, oozing, and crusting). A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by percentage of subjects with Investigator's Global Assessment score of 0 or 1 with improvement by at least 2 grades.
Time to Investigator's Global Assessment response | Within 24 Weeks
  Investigator's Global Assessment measures the severity of atopic dermatitis (0 = Clear; 1 = Almost clear; 2 = Mild disease; 3 = Moderate disease; 4 = Severe disease/Very severe disease) of clinical characteristics (erythema, infiltration, papulation, oozing, and crusting). A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by time to Investigator's Global Assessment response (Investigator's Global Assessment score of 0 or 1, with improvement by at least 2 grades).
Success rate in Eczema Area and Severity Index 50 (improvement of ≥50% in Eczema Area and Severity Index) | 24 Weeks
  Eczema Area and Severity Index measures the severity of skin symptoms. The maximum Eczema Area and Severity Index score is 72 points. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by success rate in Eczema Area and Severity Index 50 (improvement of ≥50% in Eczema Area and Severity Index).
Success rate in Eczema Area and Severity Index 75 (improvement of ≥75% in Eczema Area and Severity Index) | 24 Weeks
  Eczema Area and Severity Index measures the severity of skin symptoms. The maximum Eczema Area and Severity Index score is 72 points. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by success rate in Eczema Area and Severity Index 75 (improvement of ≥75% in Eczema Area and Severity Index).
Success rate in Eczema Area and Severity Index 90 (improvement of ≥90% in Eczema Area and Severity Index) | 24 Weeks
  Eczema Area and Severity Index measures the severity of skin symptoms. The maximum Eczema Area and Severity Index score is 72 points. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by success rate in Eczema Area and Severity Index 90 (improvement of ≥90% in Eczema Area and Severity Index).
Change from baseline in Investigator's Global Assessment | 24 Weeks
  Investigator's Global Assessment measures the severity of atopic dermatitis (0 = Clear; 1 = Almost clear; 2 = Mild disease; 3 = Moderate disease; 4 = Severe disease/Very severe disease) of clinical characteristics (erythema, infiltration, papulation, oozing, and crusting). A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by the change from baseline in Investigator's Global Assessment.
Change from baseline in the total score of Eczema Area and Severity Index and each clinical sign score | 24 Weeks
  Eczema Area and Severity Index measures the severity of skin symptoms. The maximum Eczema Area and Severity Index score is 72 points. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by change from baseline in the total score of Eczema Area and Severity Index and each clinical sign score.
Change from baseline in the total score of Patient-Oriented Eczema Measure | 24 Weeks
  Eczema will be evaluated according to Patient-Oriented Eczema Measure .The subjects will answer 7 questions and describe their eczema. The investigator will confirm their responses and record the results in the source document and CRF. The total score of POEM is 28 points at the most. A higher score represents a severer clinical impression on the patient's severity based on investigator/clinician's judgment.
  The efficacy is assessed by Change from baseline in the total score of Patient-Oriented Eczema Measure.
Change from baseline in the total affected Body Surface Area (percent) | 24 Weeks
  The efficacy is assessed by change from baseline in the total affected Body Surface Area (percent).

CONTACTS AND LOCATIONS:
Overall Officials: Lin Ma, Principal Investigator — Beijing Children's Hospital
Locations (1):
- Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No